CLINICAL TRIAL: NCT00738764
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation Trial of PDL192 in Subjects With Advanced Solid Tumors
Brief Title: A Trial of PDL192 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDL192-1801
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2011-12

CONDITIONS: Cancer
Keywords: cancer; antibody; Phase 1 Clinical Trial
MeSH Terms: conditions — Neoplasms | interventions — enavatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): PDL192 Dose Level 1
  Interventions: Biological: PDL192
- Cohort 2 (Experimental): PDL192 Dose Level 2
  Interventions: Biological: PDL192
- Cohort 3 (Experimental): PDL192 Dose Level 3
  Interventions: Biological: PDL192
- Cohort 4 (Experimental): PDL192 Dose Level 4
  Interventions: Biological: PDL192
- Cohort 5 (Experimental): PDL192 Dose Level 5
  Interventions: Biological: PDL192
- Cohort 6 (Experimental): PDL192 Dose Level 6
  Interventions: Biological: PDL192

INTERVENTIONS:
Biological: PDL192 — Humanized anti-TWEAK receptor monoclonal IgG1 antibody

SUMMARY:
This is a phase 1, multicenter, open-label, dose escalation trial of PDL192 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
The primary study objective is to determine the maximum tolerated dose of PDL192 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria

Eligible subjects will be considered for inclusion in this study if they meet all of the following criteria:

1. Male or female, 18 years of age or older.
2. Subjects with documented advanced solid tumors.
3. Subjects who have previously failed all standard therapies or subjects who have a tumor where no standard therapy exists.
4. A negative serum pregnancy test (women of childbearing potential only) at screening. Male or female subjects of reproductive potential must be willing to use adequate contraception during the duration of the study and for a minimum of 3 months after the end of treatment.
5. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Exclusion Criteria

Subjects will be ineligible for this study if they meet any one of the following criteria:

1. Symptomatic and progressive central nervous system (CNS) metastases or leptomeningeal metastases
2. Diagnosis of glioblastoma
3. Eastern Cooperative Oncology Group (ECOG) performance status >= 2
4. Abnormal hematologic values defined as:

   * Hemoglobin level < 9 g/dL
   * Absolute neutrophil count (ANC) < 1500/mm3
   * Platelet count < 100,000/mm3
5. Abnormal kidney, liver, or pancreatic function defined as:

   * Serum creatinine > 1.5 x upper limit of normal value (ULN)
   * Aspartate transaminase or alanine transaminase levels of > = 2.5 x ULN
   * Bilirubin > ULN
   * Amylase > 1.5 x ULN
   * Lipase > 1.5 x ULN
6. Known chronic viral hepatitis
7. History of cirrhotic liver disease
8. History of pancreatitis (patients with history of gall stone pancreatitis who are status post-cholecystectomy will be eligible)
9. Acute cholecystitis within 6 months prior to the first dose of study drug
10. Treatment with any investigational drug, antineoplastic agent, or antibodies within 21 days prior to the first dose of study drug (6 weeks for vaccines or nitrosureas)
11. Proteinuria >1 g/24 hours (only subjects with > = 2+ with dipstick test will undergo 24 hour urine collection)
12. Ongoing >= Grade 2 toxicities resulting from prior therapies
13. Received continuous systemic steroids at doses greater than 10 mg/day of prednisone or its equivalent within 30 days prior to the first dose of study drug (intermittent dexamethasone given for prophylaxis or treatment of emesis is permitted)
14. Received any immunosuppressive agent (except steroids) within 21 days prior to the first dose of study drug
15. Known hypersensitivity to any component of the PDL192 formulation
16. Uncontrolled medical problems such as diabetes mellitus, pancreatitis, coronary artery disease, hypertension, unstable angina, arrhythmias, pulmonary disease, or symptomatic heart failure
17. Female subjects who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | after four weeks of dosing

SECONDARY OUTCOMES:
The incidence and frequency of dose-limiting toxicities; The frequency, severity, and relationship of adverse events and serious adverse events;Incidence of abnormal findings in physical examinations and clinical laboratory values | during estimated average 4 month treatment period and 90 day follow up
Pharmacokinetic profile of PDL192 including maximum serum drug concentration, area under the concentration-time curve from time zero to infinity, systemic clearance, volume of distribution, and elimination half-life | during estimated average 4 month treatment period and 90 day follow up
Incidence of PDL192-specific antidrug antibodies | during estimated average 4 month treatment period and 90 day follow up
Objective response rate (Complete Response + Partial Response) and Disease control rate (Complete Response + Partial Response + Stable Disease) | during estimated average 4 month treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Obrocea, MD, Study Director — Abbott Biotherapeutics Corp.
Locations (2):
- United States (2):
  - Site Reference ID/Investigator# 53365, Scottsdale, Arizona
  - Site Reference ID/Investigator# 53364, Aurora, Colorado